CLINICAL TRIAL: NCT04584567
Title: Covid-19 Infection Prophylaxis With Low Dose of Doxycycline and Zinc in Health Care Workers
Brief Title: OD-doxy-PNV-COVID-19 Old Drug " DOXY " for Prevention of New Virus " COVID-19 "
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hedi Gharsallah (Network)
Collaborators: Dacima Consulting (Other)
Responsible Party: Sponsor-Investigator, Hedi Gharsallah, Professor, General Administration of Military Health, Tunisia
Organization: General Administration of Military Health, Tunisia (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UR17DN05
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: The participants who meeting study entry criteria will be randomized in a 1:1 blinded comparison of daily low dose DOXY versus oral placebo for 6 weeks.
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DOXY ZINC (Experimental): Doxycycline daily dosing (100mg) Zinc daily dosing (15mg)
  Interventions: Drug: Doxycyclin
- DOXY PLACEBO (Placebo Comparator): Doxycycline daily dosing (100mg) placebo of Zinc
  Interventions: Drug: Doxycyclin
- PLACEBO (Placebo Comparator): placebo of Doxycycline daily dosing placebo of Zinc
  Interventions: Drug: Doxycyclin

INTERVENTIONS:
Drug: Doxycyclin — daily (100mg)

SUMMARY:
Given the urgency of having guidelines for the management of COVID-19 in the current epidemic context and the lack of specific pharmacological treatment, Military Health recommends the launch of a multicenter, randomized, double-blind, interventional clinical trial.

The aim of this study is to evaluate the efficacy of a combination of two treatments, low-dose doxcycline (100 mg/day) and Zinc (15 mg/day) (dietary supplement) in the primary prevention of COVID-19 infection in health care professionals in Tunisia compared to two control groups.

ELIGIBILITY:
Inclusion Criteria:

* No self-medication with study drugs or antivirals
* Negative COVID19 diagnosis confirmed by PCR and negative Elisa antibody assay
* No signs of COVID19
* Having given consent for the study

Exclusion Criteria:

Participation in other clinical trials aimed at primary prevention of VIDOC infection19

* Liver failure
* Known allergy to the study product
* Pregnancy or breastfeeding
* Vitamin A and E treatment in progress

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
decreasing the number of cases infected with covid 19 | WEEK 6
  Determine if the use of doxyciciline low dose as preventive treatment decrease the number of cases infected with covid 19 in the active arm compared to the placebo arm. Participants for each randomized treatment arm as compared to placebo.

SECONDARY OUTCOMES:
Measurement of the emergence of clincal symptoms of COVID 19 | WEEK 6
  Comparison of the emergence of clinical symptoms or COVID-19 diagnosis in participants presenting asymptomatically at study entry but identified as seropositive by serology at entry between the randomized treatment arms and comparator arm.
the seroprevalence of SARS- CoV 2 IgM/IgG positive samples at study entry and study conclusion in all participants receiving DOXY compared to those receiving placebo. | WEEK 6
  Comparison of the rate of SARS-CoV 2 infections as measured by IgM/IgG seroconversion in study participants receiving randomized DOXY versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Batikh R Riadh, physican, Study Chair — Military hospital; Stambouli N nejla, phd, Study Director — Military hospital; Gharsallah H Hedi, physican, Principal Investigator — Military hospital; Ferjani M Mustapha, physican, Study Chair — Direction de la Santé militaire; Ben Moussa M mohamed, physican, Study Chair — Military hospital; Youssfi MA Mohamed Al, physican, Study Chair — Military hospital
Locations (1):
- Military Hospital of Tunis, Tunis, Montfleury, Tunisia

IPD SHARING:
Plan to Share IPD: No